CLINICAL TRIAL: NCT04393701
Title: A Pilot Study for Systematic Neonatal Screening for Lysosomal Storage Diseases Using Tandem Mass Spectrometry
Acronym: LysoNeo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Collaborators: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020/0007/HP
Record Dates: First submitted 2020-05-14; First posted 2020-05-19 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Neonatal Screening; Lysosomal Storage Diseases
MeSH Terms: conditions — Lysosomal Storage Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- neonates tested in Normandie, France (Experimental): All neonates will be tested in Normandie
  Interventions: Procedure: Additional blood sampling

INTERVENTIONS:
Procedure: Additional blood sampling — Additional blood sampling on blotting paper will be done in neonates in Normandy, France, compared to National neonatal screening program

SUMMARY:
The study will include all newborns in Normandie region for 3 years (about 105,000 births) for whom signed consent by one (or two) parents will be collected. Based on our previous pilot study (2011) assessing MCAD and PKU using tandem mass spectrometry-based method in Normandie region in which informed consents have been signed for all newborns (43,000) but we are expecting a great willingness to participate to this project. Thus, we are aiming to include 100,000 newborns, and the study will be continued until we reach at least this target.

The primary objective is to evaluate the epidemiology of MPS1 and Pompe disease using dried blood samples in the first cohort of neonates tested in France (Normandie region).

ELIGIBILITY:
Inclusion Criteria:

* Newborn in a Normandy maternity hospital
* Newborn participating in the National Neonatal Screening Program
* Holder(s) of parental authority having read and understood the information letter and signed the informed consent form

Exclusion Criteria:

There are no criteria for non-inclusion in this study. Participation in the study, such as participation in the National Neonatal Screening Program, is not mandatory.

Ages: 1 Day to 4 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100000 (Estimated)
Dates: Start 2021-03-08 (Actual); Primary Completion 2026-12-08 (Estimated); Study Completion 2026-12-08 (Estimated)

PRIMARY OUTCOMES:
Number of newborns in relation to the number of cases of blotting paper collected | From day 2 to day 4

SECONDARY OUTCOMES:
Number of newborns with positive sample for Mucopolysaccharidosis type I | From day 2 to day 4
Number of newborns with positive sample for Pompe disease | From day 2 to day 4

CONTACTS AND LOCATIONS:
Overall Officials: Soumeya BEKRI, Pr, Principal Investigator — University Hospital, Rouen
Locations (2):
- France (2):
  - Caen University Hospital, Caen
  - Rouen University Hospital, Rouen

IPD SHARING:
Plan to Share IPD: No